CLINICAL TRIAL: NCT05741801
Title: Digital Alerting to Improve Sepsis Detection and Patient Outcomes in NHS Trusts. A Qualitative Study (DiAlS Qual).
Brief Title: Digital Alerts for Sepsis: a Qualitative Study
Acronym: DiAlSQual
Status: Completed | Type: Observational
Sponsor: University of Oxford (Other)
Collaborators: Institute of Cancer Research, United Kingdom (Other)
Responsible Party: Sponsor
Other Study IDs: 16347
Record Dates: First submitted 2023-01-31; First posted 2023-02-23 (Actual); Last update posted 2024-08-28 (Actual); Status verified 2023-01

CONDITIONS: Sepsis
Keywords: digital alerts; NHS England hospitals; emergency departments; electronic patients records; outreach teams; decision support systems; patient deterioration scores; antibiotics administration
MeSH Terms: conditions — Sepsis; Emergencies | interventions — Interviews as Topic; Focus Groups; Watchful Waiting

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- health care professionals: Hospital healthcare professionals who use, or help implement, deteriorating patient/sepsis alerts in NHS trusts.
  Interventions: Other: interviews
- ex-patients/survivors and family members/carers: Ex-patients recruited from NHS trusts and other charities, who have previously had sepsis or family members of patients who have had sepsis.
  Interventions: Other: interviews

INTERVENTIONS:
Other: interviews — observations of healthcare professionals working in hospitals (outreach/sepsis team), one-on-one interviews with healthcare professionals, and focus groups or interviews with ex-patients/family members.
  Other Names: focus groups; observations

SUMMARY:
Sepsis is a serious disease, most often caused by a bacterial infection, and can be treated with antibiotics. Identifying patients with sepsis as early as possible means treatment with antibiotics can be started earlier. To identify patients who may have sepsis, measurements such as high or low temperature and fast breathing rate are used to create a score showing the possibility of sepsis. Electronic Health Records (EHRs) in hospitals contain the information needed to create a score and can alert a doctor or nurse that a patient may have sepsis. Research has shown that more patients get antibiotics earlier because of hospitals using this type of digital alert. Different hospitals have used different methods to create a score and use different types of digital alerts. This research wants to find out what hospital doctors and nurses think about digital alerts for sepsis and how they use them. The investigators also want to find out what patients who have had sepsis think about hospitals using these digital alerts. Understanding how these digital alerts are used and how they affect patient care can help see how they could be used better so patients can benefit.

DETAILED DESCRIPTION:
Sepsis is a common cause of serious illness and death with an estimated 123,000 cases and 46,000 deaths in the UK each year. Similarly, high levels of sepsis have been reported internationally, and sepsis is recognised by the World Health Organisation as a global health priority. Many countries have nationwide sepsis action plans and all UK hospitals have set targets to rapidly diagnose and treat patients with sepsis. Timely appropriately targeted intravenous antibiotics have been shown to be effective in improving outcomes for patients, with a 4% increase in odds of mortality for every hour's delay in administration of intravenous antibiotics.

The need for rapid treatment has led to the development of clinical criteria and 'screening tools' have been proposed to identify patients with sepsis. These include Sequential (Sepsis related) Organ Failure Assessment (Sofa), Systemic Inflammatory Response Syndrome (SIRS) criteria and in England the National Early Warning Score (NEWS), which was developed by the UK Royal College of Physicians. In December 2017, an updated version of NEWS, NEWS2 was published, which is recommended by NICE and the Royal College of Physicians as the most effective screening tool for sepsis in the UK. Available tools are based on current observations which clinicians are able to take and quickly calculate a score, but there is a paucity of evidence as to which tool to use and their effect on patient outcomes.

Potential pathways for the effectiveness of alerts when clinical deterioration is due to sepsis are likely to include an increase in the proportion of patients receiving intravenous antibiotics in one hour, and other 'sepsis six' measures. Improved communication and changes in dialogue between healthcare teams has been suggested as an important pathway for improvements in clinical outcomes. In addition, the introduction of sepsis alerts is often accompanied by treatment plans as well as education and training activities. Little is known about the contribution of these and other potential mediators on the effectiveness of alerts.

Previous qualitative research with healthcare professionals has highlighted problems in identification and management of sepsis including limits in professionals' capacity to identify sepsis, difficulties in handover of patients and errors in communication. These studies highlight both the requirement for healthcare professionals to feel confident in their assessment of patients and for clinical and organisations structures to work efficiently to provide optimal patient care. Previous qualitative research with patients has reported on patients' decisions to seek help with symptoms, experiences of hospitalisation and how patients have managed life after surviving sepsis. Additional studies with caregivers have described the burden on those caring for sepsis survivors and their role in advocating for their loved ones. Another study has looked at the words patients and call handlers use to describe symptoms of sepsis when patients seek help. These topics can help inform how patients and clinicians could use and potentially benefit from the use of digital alerts in hospitals.

This study is part of a wider programme of work seeking to determine the effectiveness of the introduction of digital alerts to improve outcomes of patients with sepsis. This component of the work seeks to explore healthcare professionals' and patients'/family members' views and experiences of deteriorating patient/sepsis alert systems in hospitals. This work will be undertaken within at least some of the NHS Trusts involved in the wider programme of work (Royal Berkshire NHS Foundation Trust, Oxford University Hospitals NHS Foundation Trust, University College London Hospitals NHS Foundation Trust, Imperial College Healthcare NHS Trust, Chelsea and Westminster Hospital NHS Foundation Trust and Cardiff & Vale University Health Board) and potentially additional Trusts if required.

This is a qualitative study which includes three methods of data collection; observation of healthcare professionals working in hospitals, one-to-one interviews with healthcare professionals and interviews/focus groups with patients/family members.

Healthcare professionals will include doctors, nurses and other professionals who use, or help implement, deteriorating patient/sepsis alerts in NHS hospital Trusts. Patients/family members will include patients recruited from NHS trusts and community settings, who have previously had sepsis or are family members of patients who have had sepsis.

Interviews and focus groups will include topics which may be upsetting for some patients/family members or healthcare professionals. All participants will be made aware of sources of support available to them through the NHS and other relevant organisations. Patients and family members will have the option of taking part in a focus group or an individual interview depending on what they feel comfortable with.

ELIGIBILITY:
Inclusion Criteria:

* Healthcare Professionals

  * Participant is willing and able to give informed consent for participation in the study.
  * Any gender aged 18 years or above (no upper age limit).
  * Fluent in English (or able to participate in an interview with other measures in place, e.g. interpreter).
  * Currently working as a healthcare professional (e.g. doctor, nurse) in an NHS hospital trust.

Ex-Patients and Family Member

* Participant is willing and able to give informed consent for participation in the study.
* Any gender aged 18 years or above (no upper age limit).
* Fluent in English (or able to participate in an interview with other measures in place, e.g. interpreter).
* Member of the public who has previously been diagnosed with sepsis and treated in hospital or family member/carer of someone who has previously had sepsis.

Exclusion Criteria:

* The participant may not enter the study if ANY of the following apply:

  * Healthcare professional has less than 3 months experience working in relevant role. This is estimated to be a reasonable amount of time for them to have good experience of identifying patients with sepsis and/or using sepsis alert systems.

Ages: 18 Years to 80 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Participants will include hospital healthcare professionals and ex-patients/family members in the UK.
  The sample size will depend on saturation, i.e. no new themes are identified in data from later interviews/focus groups, however it is estimated that around 30 healthcare professionals and 20 patients/family members will participate.
  Analysis of data from the interviews and the focus groups will occur concurrently to data collection, where possible, to inform future sampling and data collection.
Sampling Method: Non-Probability Sample
Enrollment: 39 (Actual)
Dates: Start 2022-11-04 (Actual); Primary Completion 2023-07-17 (Actual); Study Completion 2023-07-17 (Actual)

PRIMARY OUTCOMES:
In-depth, one-to-one, semi-structured interviews [or focus groups] on views and experience on sepsis digital alerts | June 2023
  The views and experiences of healthcare professionals and patients/family members on sepsis/deteriorating patient alert systems in hospitals is analysed, as well as on general identification and management of sepsis.

SECONDARY OUTCOMES:
Observations on use on sepsis digital alerts within the hospital digital system | June 2023
  1. To understand how healthcare professionals use sepsis alerts and how alerts influence their decision making.
  2. To observe healthcare professionals use of sepsis alerts during routine hospital shifts.
  3. To identify barriers and facilitators to the implementation and use of digital sepsis alerts in NHS hospital settings.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Oxford, Oxford, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Lazzarino R, Borek AJ, Brent AJ, Welch J, Honeyford K, Daniels R, Kinderlerer A, Cooke G, Patil S, Gordon A, Goodman P, Glampson B, Ghazal P, Costelloe C, Tonkin-Crine S. The sepsis journey and where digital alerts can help: a qualitative, interview study with survivors and family members in England. Front Public Health. 2025 Mar 26;13:1521761. doi: 10.3389/fpubh.2025.1521761. eCollection 2025. PMID 40231176